CLINICAL TRIAL: NCT00697476
Title: Phase I-II Study of Oral Suberoylanilide Hydroxamic Acid (Vorinostat) in Combination With Topotecan in Patients With Chemosensitive Recurrent Small Cell Lung Cancer (SCLC)
Brief Title: Study of Oral Vorinostat in Combination With Topotecan in Patients With Chemosensitive Recurrent SCLC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, MD, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2007-002; 2008-002125-37 (EudraCT Number)
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Small Cell Lung Cancer
Keywords: second line chemotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vorinostat/Topotecan (Experimental): Vorinostat/topotecan dose escalation regimen. vorinostat is administered orally once a day for 7 to 14 consecutive days, according to the dose level.Topotecan is administered I.V. for 5 consecutive days every three weeks.
  Vorinostat dose levels go from 300 mg/day for 7 days to 400 mg/day for 14 days. Topotecan dose levels go from 1,2 mg/m2 to 1,5 mg/m2
  Interventions: Drug: topotecan, vorinostat

INTERVENTIONS:
Drug: topotecan, vorinostat — Phase I study: vorinostat will be administered daily for a number of days per cycle variable from 7 to 14 according to the level of dose escalation; topotecan will be administered I.V. for 5 consecutive days every 3 weeks.
  Phase II study: Patients will receive treatment at the recommended dose established by phase I part of the trial, for a maximum of 6 cycles or until disease progression, unacceptable toxicity or patient's refusal.
  Other Names: Merck Vorinostat

SUMMARY:
The purpose of this study is to evaluate the maximum tolerated dose, the activity and the safety profile of the combination of vorinostat and topotecan in patients with recurrent small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of SCLC;
* Limited or extensive-stage disease in patients who have received a single chemotherapy regimen or combined modality (chemotherapy + chest radiotherapy) regimen and relapsed after completion of first-line chemotherapy (sensitive relapse);
* Age >/= 18 years;
* ECOG Performance Status 0-2;
* Life expectancy of at least 12 weeks;
* Measurable lesions according to RECIST criteria;
* Adequate cardiac, hepatic, renal, and bone marrow function;
* Written informed consent.

Exclusion Criteria:

* Prior treatment with an HDAC inhibitor;
* Symptomatic and/or unstable pre-existing brain metastases;
* Superior Vena Cava Syndrome;
* Spinal cord compression;
* Severe or uncontrolled medical diseases (Hypertension, diabetes, congestive heart failure, myocardial infarction within 6 months of study, chronic renal disease, or active uncontrolled infections);
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ;
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of the combination as the recommended dose for phase II trial [Phase I]; objective response rate of the combination [Phase II]; toxicity and safety profile of the combination [Phase II] | Limiting tolerated dose (Phase I); efficacy/toxicity after the inclusion of the last patient (Phase II)

SECONDARY OUTCOMES:
To assess the antitumor activity of the combination in terms of time to progression (TTP) and overall survival (OS) [Phase II] | After the follow up period

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy